CLINICAL TRIAL: NCT00723385
Title: Effects of Vitamin D on Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AG0104; 5R01AG015982 (NIH)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia; Vitamin D Deficiency
Keywords: cholesterol; LDL-cholesterol; cholecalciferol; lipids; C-reactive protein
MeSH Terms: conditions — Hypercholesterolemia; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administration for 12 weeks with repeated 25-OH D determinations over 12 weeks, dietary, sunshine questionnaire recording
  Interventions: Other: Placebo
- Vitamin D (Experimental): Vitamin D (1000 or 2000 IU/day)
  Interventions: Dietary Supplement: Vitamin D (1000 or 2000 IU/day)

INTERVENTIONS:
Dietary Supplement: Vitamin D (1000 or 2000 IU/day) — Dose titration beginning with 1000 IU/day and either remaining at 1000 IU/day for weeks 7-12 if normalized D levels at 6 weeks or increasing to 2000 IU/day for weeks 7-12 if levels not normalized at week 6
  Other Names: cholecalciferol
  Arms: Vitamin D
Other: Placebo — Administration of placebo for 12 weeks with repeated D measurements
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether oral vitamin D supplementation in people with inadequate vitamin D concentrations will lower LDL-cholesterol and total cholesterol concentrations.

DETAILED DESCRIPTION:
Data from previous trials suggest a protective role of vitamin D in cardiovascular disease. A recent meta-analysis of trials with at least 5 years of follow-up of vitamin D supplementation concluded that intake of vitamin D supplements may decrease total mortality, but that the relationship between baseline vitamin D status, dose of vitamin D supplements, and total mortality rates remains to be investigated. An even more recent analysis of vitamin D concentrations found that participants with vitamin D deficiency and hypertension were about twice as likely as people without hypertension and vitamin D deficiency to have a cardiovascular event during the study.

The main hypothesis to be tested is that normalization of vitamin D levels will lower LDL-cholesterol and total cholesterol concentrations in people with inadequate vitamin D concentrations as determined by circulating 25-OH vitamin D. Subhypotheses are that HDL-cholesterol, triglycerides, lipoprotein(a), hs C-reactive protein and Hemoglobin A1c will not be affected, and that cyp3a-metabolized medication levels will decrease with vitamin D replacement.

This is a 12-week randomized double-blind dose titration study of the effects of supplementation with 1000-2000 IU vitamin D on lipid and vitamin D concentrations. Dietary intake of vitamin D will be estimated by dietary recall questionnaire or analysis of three non-consecutive 24-hour dietary intake logs.

ELIGIBILITY:
Inclusion Criteria:

* Any medically stable person able to swallow pills
* Inadequate vitamin D status at screening visit

Exclusion Criteria:

* Clinical instability of underlying disease process (e.g., recent hospitalization, change of dosages of medications within the prior two weeks, or new medications within one month)
* Recent transfusion
* Severe renal failure or dialysis
* Hypercalcemia
* Malignancy under active treatment
* Feeding tube
* Intestinal bypass surgery
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | 12 weeks

SECONDARY OUTCOMES:
Vitamin D and metabolite concentrations with supplementation and time course of repletion in deficient or insufficient subjects | 12 weeks
Measures of inflammatory markers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janice B. Schwartz, MD,FACC,FAHA, Principal Investigator — Jewish Home, University of California, San Francisco
Locations (1):
- Jewish Home, San Francisco, California, United States

REFERENCES:
- [Background] Autier P, Gandini S. Vitamin D supplementation and total mortality: a meta-analysis of randomized controlled trials. Arch Intern Med. 2007 Sep 10;167(16):1730-7. doi: 10.1001/archinte.167.16.1730. PMID 17846391
- [Background] Wang TJ, Pencina MJ, Booth SL, Jacques PF, Ingelsson E, Lanier K, Benjamin EJ, D'Agostino RB, Wolf M, Vasan RS. Vitamin D deficiency and risk of cardiovascular disease. Circulation. 2008 Jan 29;117(4):503-11. doi: 10.1161/CIRCULATIONAHA.107.706127. Epub 2008 Jan 7. PMID 18180395
- [Result] Kane L, Moore K, Lutjohann D, Bikle D, Schwartz JB. Vitamin D3 effects on lipids differ in statin and non-statin-treated humans: superiority of free 25-OH D levels in detecting relationships. J Clin Endocrinol Metab. 2013 Nov;98(11):4400-9. doi: 10.1210/jc.2013-1922. Epub 2013 Sep 12. PMID 24030939